CLINICAL TRIAL: NCT00633113
Title: A Randomized, Prospective, Blinded Clinical Trial Comparing Two Total Knee Replacement Techniques
Brief Title: Minimally Invasive Knee Replacement Outcomes (MIKRO) Study
Acronym: MIKRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MIKRO
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Minimally Invasive Knee Replacement; Knee Osteoarthritis; Cost effectiveness minimally invasive knee surgery
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — 15-phenyl-beta-methylpentadecanoic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): - Medial Parapatellar Arthrotomy (MPPA) technique
  Interventions: Procedure: MPPA
- 2 (Active Comparator): - Subvastus (SV) technique
  Interventions: Procedure: SV

INTERVENTIONS:
Procedure: MPPA — - Medial Parapatellar Arthrotomy
  Arms: 1
Procedure: SV — - Subvastus Technique
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate and compare the clinical, radiographic (x-ray) and cost effectiveness outcomes (cost relative to risks and benefits) of two different minimally invasive knee joint replacement surgical techniques. The primary study hypothesis is that in comparing total knee replacement performed with the two different surgical techniques that respect four minimally invasive surgery principles (low-profile instrumentation, "minimally invasive" incision, overall minimal knee surgical intervention), a faster return to function will result when the technique does not incise the tendon.

DETAILED DESCRIPTION:
This study does not include financial compensation for treatments involved.

ELIGIBILITY:
Inclusion Criteria:

* Presence of severely symptomatic knee osteoarthritis that has failed non- operative treatment
* Males and non-pregnant females, 35-85 years of age at the time of surgery
* ASA class 1 or 2
* Procedure will not require computer navigation
* Patient/Surgeon has not requested another implant
* Patient has signed an IRB approved study consent form
* Patient is able and willing to actively participate in post-operative rehabilitation program
* Patient understands study requirements
* Patient is willing to comply with follow-up visits and diary documentations
* Patient is capable of independent ambulation

Exclusion Criteria:

* Skeletal immaturity
* More than 10 degrees of valgus or varus deformity as measured from a weight bearing AP alignment view
* Patients with bilateral knee osteoarthritis who are considering a simultaneous bilateral procedure
* Bone or ligament insufficiency that requires the use of augments or stems, or constrained component
* Daily pre-operative use of narcotic pain medication
* Prior knee arthroplasty
* Patient is a prisoner
* Patient has had prior tibial tubercle osteotomy
* Patient's surgical knee would require removal of hardware prior to TKA
* Patient has < 95 degrees flexion pre-operatively

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome: clinical outcomes in the Subvastus Total Knee Arthroplasty versus Medial Parapatellar surgical groups, using the Knee Society Score. | 5 years

SECONDARY OUTCOMES:
Secondary outcome: Includes cost-effectiveness of the Subvastus Total Knee Arthroplasty versus Medial Parapatellar surgical groups; EQ-5D, SF-12; radiographic assessment using Knee Society Radiographic Assessment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ivan M Tomek, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States